CLINICAL TRIAL: NCT06846853
Title: Gadopiclenol vs. Gadobutrol for Dynamic Contrast-Enhanced Pituitary MRI: A Pilot Study
Brief Title: Gadopiclenol vs. Gadobutrol for Dynamic Contrast-Enhanced Pituitary MRI (Magnetic Resonance Imaging)
Acronym: MRI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Leo Wolansky, Professor, UConn Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 25-175-1
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Contrast Enhanced Images vs. Non-contrast Images; Gadopiclinol Enhanced Images vs. Gadobutrol Enhanced Images
Keywords: Gadobutrol enhanced images; Gadopiclinol enhanced images
MeSH Terms: interventions — gadopiclenol; gadobutrol

STUDY DESIGN:
Intervention Model Description: This is a double-blinded cross-over study. Study participants will be assigned randomly to have either Gadopiclenol or Gadobutrol contrast for the first MRI scan and followed by the other contract for the second MRI scan 3-14 days later.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gadopiclinol (brand name, Elucirem) first group (Experimental): Participants of Arm 1 will use Gadopiclinol (Brand name, Elucirem) contrast for the first MRI scan and use Gadobutrol (Brand name, Gadavist)contrast for the second MRI scan
  Interventions: Drug: Gadopiclenol
- Gadobutrol (Brand name, Gadavist) first group (Active Comparator): Participants of Arm 2 will use Gadobutrol contrast for the MRI scan and Gadopiclinol contrast for the second MRI scan.
  Interventions: Drug: Gadobutrol (Gadavist, BAY86-4875)

INTERVENTIONS:
Drug: Gadopiclenol — The enhanced images by Gadopiclenol and Gadobutrol will be compared.
  Arms: Gadopiclinol (brand name, Elucirem) first group
Drug: Gadobutrol (Gadavist, BAY86-4875) — Gadobutrol will be used as a comparator
  Arms: Gadobutrol (Brand name, Gadavist) first group

SUMMARY:
This study will evaluate the efficacy and safety of Gadopiclenol, an FDA-approved contrast agent, for visualizing pituitary lesions on MR images by comparing with the comparator, Gadobutrol, a clinically widely used contrast agent. The study is double-blinded, so neither the participants nor the researchers know which contrast agent is being used during each scan to avoid the bias of results.

DETAILED DESCRIPTION:
Gadopiclenol (brand name Elucirem), initially invented by Guerbet, is an FDA-approved macrocyclic gadolinium-based contrast agent (GBCA) with high relaxivity and high kinetic stability. The higher relaxivity allows for a lower dose of gadopiclenol, reducing the total amount of gadolinium administration (hence reducing the toxicity of gadolinium) while preserving imaging quality.

Gadopiclenol was approved by the FDA with a recommended dose of 0.05 mmol/kg for adults and pediatric patients aged 2 years and older. The PICTURE Trial demonstrated that Gadopiclenol at 0.05 mmol/kg which is half dose of standard macrocyclic GBCAs (Gadobutrol at 0.1 mmol/kg) revealed noninferiority for contrast-enhancing intracranial lesions against the background of nonenhancing brain.

A pituitary microadenoma or a Rathke's cyst is typically demonstrated on MRI by virtue of hypoenhancement of the lesion against the background of the hyperenhancing pituitary. Dynamic pituitary imaging with Gadopiclenol has not been investigated so far.

This pilot study will assess the value of Gadopiclenol at 0.05 mmol/kg vs. Gadobutrol 0.1 mmol/kg as a contrast agent for MRI in the evaluation of pituitary lesions. We hypothesize that there will be a trend that Gadopiclenol will increase the enhancement of the background pituitary gland to a similar degree. The safety data utilizing Gadopiclenol will also be evaluated. We anticipate comparable safety of 0.05 mmol/kg of Gadopiclenol and 0.1 mmol/kg Gadobutrol.

ELIGIBILITY:
Inclusion criteria:

1. Male adult patient who is at 18 years old or above, or female adult patient who is at 55 years old or above.
2. Patient presenting with known or highly suspected pituitary lesion(s) with focal areas of disrupted Blood Brain Barrier (BBB) (e.g., primary and secondary tumors) based on results of a previous imaging procedure such as Computed Tomography (CT) or MRI, which should have been performed within 12 months prior to informed consent form signature.
3. Patient scheduled for a contrast-enhanced MRI examination with a focus on pituitary for clinical reasons and agreeing to have a second contrast-enhanced MRI examination for the purpose of the trial.
4. If the patient was treated (either with radiation, surgery, biopsy or other relevant treatments) for a pituitary condition between previous imaging evaluation and trial MRI, there should still be a high suspicion of remaining lesion(s) on the basis of available clinical information.
5. Patient able and willing to participate in the trial.
6. Patient having read the information and having provided his/her consent to participate in writing by dating and signing the informed consent prior to any trial related procedure being conducted.
7. Patient affiliated to national health insurance according to local regulatory requirements.

Exclusion criteria:

1. Patient presenting with known class III/IV congestive heart failure according to the New York Heart Association classification (NYHA).
2. Patient having received any investigational medicinal product within 7 days prior to trial entry or scheduled to receive any investigational treatment in the course of the trial.
3. Patient presenting with any contraindication to MRI examinations.
4. Patient previously randomized in this trial.
5. Patient having received any contrast agent (MRI or CT) within 3 days prior to first trial product administration, or scheduled to receive any contrast agent during the course of the trial or within 24 hours after the second trial product administration
6. Patient expected/scheduled to have any treatment or medical procedure (e.g. chemotherapy, radiotherapy, biopsy or surgery etc.) that may impact the aspects of the imaged lesions between the 2 MRI examinations. (Patients under corticosteroids and/or maintenance chemotherapy with a stable dose at the time of screening visit and throughout the trial can be included).

Patient with anticipated, current or past condition (medical, psychological, social or geographical) that would compromise the patient's safety or her/his ability to participate in the trial.

8. Patient unlikely to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits and/or unlikelihood of completing the trial.

9. Patient related to the investigator or any other trial staff or relative directly involved in the trial conduct. 10. Patient presenting with acute or chronic renal insufficiency, defined as an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m² assessed within 1 day prior to each contrast agent injection. 11. Patient with known contra-indication(s) to the use or with known sensitivity to one of the products under investigation or to other GBCAs (such as hypersensitivity, post contrast acute kidney injury).

12. Patient who are prisoners, pregnant women, or educationally disadvantaged persons known as vulnerable population will be excluded as well to protect the rights and welfare of these participants.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
hypointense for lesions with respect to pituitary | Two MRI scans will be conducted separated by 3-14 days.
  The primary outcome measures will include both subjective assessments and an objective measure.
  The subjective assessments will include part 1) the lesion intensity of the pituitary either having: a) Not Hypointense; b) Mildly Hypointense; c) Markedly Hypointense and part 2) the overall diagnostic quality of the contrast vs noncontrast and of the two contrast agent ( Godopiclinol vs. Godobutrol) side by side as: a) Prefer 1; b) No difference; c) Prefer 2.
  The objective measure is the Contrast/Noise intensity of the pituitary:
  [Signal Intensity Background Pituitary - Signal Intensity Lesion] / Signal Intensity Air

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This study aimed to demonstrate that contrast-enhanced MRI of the central nervous system (CNS) with gadopiclenol at 0.05 mmol/kg is not inferior to gadobutrol at 0.1 mmol/kg, and superior to unenhanced MRI. The results supported the hypothesis. — https://pmc.ncbi.nlm.nih.gov/articles/PMC10090311